CLINICAL TRIAL: NCT01652937
Title: A Phase 2a, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of BIIB057 in Subjects With Rheumatoid Arthritis Who Have Had an Inadequate Response to Disease-Modifying Antirheumatic Drugs
Brief Title: BIIB057 in Subjects With Rheumatoid Arthritis and Inadequate Response to Disease-Modifying Antirheumatic Drugs
Acronym: EMBRACE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 227RA201
Record Dates: First submitted 2012-07-19; First posted 2012-07-30 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2012-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; DMARD-IR
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo + Background Therapy (Placebo Comparator): Background therapy including DMARD(s) approved by protocol
  Interventions: Drug: Placebo
- BIIB057 Dose 1 + Background Therapy (Experimental): Background therapy including DMARD(s) approved by protocol
  Interventions: Drug: BIIB057
- BIIB057 Dose 2 + Background Therapy (Experimental): Background therapy including DMARD(s) approved by protocol
  Interventions: Drug: BIIB057
- BIIB057 Dose 3 + Background Therapy (Experimental): Background therapy including DMARD(s) approved by protocol
  Interventions: Drug: BIIB057

INTERVENTIONS:
Drug: BIIB057 — Oral
  Arms: BIIB057 Dose 1 + Background Therapy; BIIB057 Dose 2 + Background Therapy; BIIB057 Dose 3 + Background Therapy
Drug: Placebo — Oral
  Arms: Placebo + Background Therapy

SUMMARY:
Phase II study designed to evaluate the safety and efficacy of BIIB057 in Subjects with Rheumatoid Arthritis who have experienced an Inadequate Response to Disease-Modifying Antirheumatic Drugs (DMARDs).

ELIGIBILITY:
Inclusion Criteria:

* Adult onset RA satisfying 2010 Revised ACR Criteria for the Classification of RA with a disease history of at least 6 months
* Active RA as defined by: at least 4 swollen joints (based on 28-joint count), at least 4 tender joints (based on 28-joint count), and high-sensitivity CRP (hsCRP) 10mg/L or greater
* No prior treatment with biologics
* Receiving a DMARD therapy for at least 3 months, using a regimen that has been stable for at least 28 days prior to screening

Exclusion Criteria:

* History of inflammatory joint disease other than RA
* Abnormal chest X-ray consistent with tuberculosis, malignancy, or infection
* History of malignancy, carcinoma in situ, or high-grade dysplasia
* History of opportunistic infection, infection requiring treatment, serious local infection, recent fever, active herpes zoster or Epstein-Barr virus, or diagnosis or family history of Creutzfeldt-Jakob disease.
* Clinically significant cardiac disease
* Treatment with prednisone >10 mg orally daily
* Intra-articular steroid injection within 28 days before screening
* Clinically significant abnormality in hematology or blood chemistry values at screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving an ACR20 response (ACR20 = American College of Rheumatology 20% response criteria change from baseline) | Week 12

SECONDARY OUTCOMES:
Assess the safety and tolerability of BIIB057 by measuring the incidence of AEs, SAEs and changes in laboratory test results during the study | Up to 16 weeks
Proportion of subjects with 28-joint count Disease Activity Score with C-reactive protein (DAS28-CRP) <3.2, <2.6, and <2.32 | Week 12
Proportion of subjects achieving ACR50 and ACR70 response | Week 12

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Quispamsis, New Brunswick
  - Research Site, Toronto, Ontario